CLINICAL TRIAL: NCT02638389
Title: Phase III Multicentric Study Evaluating the Efficacy and Safety of Sirolimus in Vascular Anomalies That Are Refractory to Standard Care
Brief Title: Efficacy and Safety of Sirolimus in Vascular Anomalies That Are Refractory to Standard Care
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VASE
Record Dates: First submitted 2015-12-09; First posted 2015-12-23 (Estimated); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Vascular Malformations
MeSH Terms: conditions — Vascular Malformations | interventions — Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with vascular malformations (Experimental): Patients with venous, lympathic or complex vascular malformations (KTS, PTEN, etc.) will receive sirolimus after completion of inclusion criteria
  Interventions: Drug: Sirolimus

INTERVENTIONS:
Drug: Sirolimus — evaluate the efficacy and safety of sirolimus in these patients
  Other Names: Rapamycine

SUMMARY:
The phosphatidylinositol 3-kinase (PI3Kinase)/Protein Kinase B (AKT)/mammalian target of rapamycin (mTor) pathway plays a role on the development and the venous/lymphatic vascular organisations.

The investigators want to study the efficacy and the safety of Rapamycin, an mTor inhibitor.

DETAILED DESCRIPTION:
The complex vascular malformations induce chronical pains and organic dysfunctions causing significant morbidity and mortality. Therefore, the investigators need to establish guidelines in order to treat these pathologies. Standard treatments such as surgery or interventional radiology are of limited efficacy and related to a high level of recurrences as well as complications. Recent preclinical studies have shown the important role of the PI3Kinase/AKT/mTor pathway on the development and the venous/lymphatic vascular organisations suggesting an appealing therapeutic target to treat patients with venous, lympathic or complex vascular malformations.

Investigators will realize a multicentric phase III study enrolling a higher number of patients to statistically evaluate the efficacy and the safety of the Rapamycin, an mTOR inhibitor, in the treatment of children and adults with vascular malformations for which conventional therapies such as surgery or sclerotherapy are ineffective or associated with high risk of important complications. Nearly 250 patients (200 adults and 50 children) will be enrolled in several european centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex vascular anomalies that are refractory to standard care such as medical treatment, surgical resection and/or sclerotherapy/embolization (ineffective or accompanied by major complications)
* Patients must have adequate medullary function: Hemoglobine> 10,0 g/dl, neutrophils >1500/mm³ and platelets > 100.000/mm³
* Patients must have the following laboratory values:
* Total serum bilirubin ≤ 1.5 x ULN (or totally bilirubin ≤ 3 x ULN with direct bilirubin ≤ 1.5 x ULN in patients with well documented Gilbert Syndrome)
* Serum alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 x ULN (or < 5.0 x ULN if hepatic metastases are present)
* Serum creatinine 1.5 x ULN. If the serum creatinine is ≥ 1.5 x ULN, then a 24-hour Creatinine Clearance must be conducted and the result must be ≥ 60 mL/min.
* Karnofsky > 50
* Patients have to be able to sign the informed consent
* Women in age of procreation have to be informed that contraceptive methods are mandatory during the study time

Exclusion Criteria:

* Any of the following concurrent severe and/or uncontrolled medical conditions, which could compromise participation in the study or interfere with the study results:
* Impaired cardiac function or clinically significant cardiac diseases, including unstable angina pectoris, ventricular arrhythmia, valvular disease with documented compromise in cardiac function, myocardial infarction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function, history of documented congestive heart failure (New York Heart Association functional classification III-IV), documented cardiomyopathy, family history of congenital long or short QT, or known history of QT/QTc prolongation of Torsades de Pointes (TdP)
* Impairment of Gastro-Intestinal (GI) function or GI disease that may significantly alter the absorption of sirolimus (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea ≥ Grade 2, malabsorption syndrome, or small bowel resection)
* Known hypersensitivity to drugs or metabolites from similar classes as study treatment.
* Patient has other concurrent severe and /or uncontrolled medical condition that would,in the investigator's judgment, contraindicated participation in the clinical study (e.g. acute or chronic pancreatitis, liver cirrhosis, active chronic hepatitis, severely impaired lung function with a spirometry ≤ 50% of the normal predicted value and/or O2 saturation ≤ 88% at rest, etc.)
* Immunocompromised patients, including known seropositivity for HIV
* Pregnant or lactating women
* Prior treatment with PI3K and/or mTOR inhibitors

Ages: 3 Months to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2016-01-25 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2030-04-01 (Estimated)

PRIMARY OUTCOMES:
Self-assesment (or parent assesment), using visual anagogic scale (0-10) of efficacy of sirolimus | every 3 months, up to 2-year period.
  * Global treatment efficacy
  * Pain
  * Local complications/symptoms (bleeding, skin tension, esthetic and functional impairment)

SECONDARY OUTCOMES:
Number of enrolled patients with treatment-related adverse events as assessed by CTCAE v4.0 | every month during the first three months and then every three months for a 2-year-treatment period
Self assessment of quality of life change induced by sirolimus | every 3 months, up to 2-year period.
  Measured by quality of life questionnaire (adapted to MOS SF-36 survey).
Volumetric changes of the malformation on sirolimus, based on magnetic resonance imaging (MRI) 12 months after sirolimus onset. | At 12 month
  Relative change of volume of the vascular malformation between the baseline MRI (before sirolimus onset) and the 12-month MRI (during sirolimus treatment)
Efficacy of sirolimus | every three months, up to 2-year period
  Change in plasma levels fibrinogen and/ or D-dimers, reflecting improvement in an abnormal intravascular coagulation consumption
Efficacy of sirolimus measured on digital photographs | every three months, up to 2-year period
  Qualitative assessment of efficacy on digital photographs

CONTACTS AND LOCATIONS:
Overall Officials: Laurence M Boon, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (3):
- Cliniques Universitaires Saint-Luc, Université Catholique de Louvain Bruxelles, Brussels, Brussels Capital, Belgium
- CHU Caen, Caen, Brittany Region, France
- Universitätsklinikum Freiburg, Freiburg im Breisgau, Germany

REFERENCES:
- [Derived] Seront E, Damme AV, Coulie J, Vikkula M, Boon LM. Personalized sirolimus regimen for vascular malformations: a retrospective analysis of VASE cohort. Orphanet J Rare Dis. 2025 Dec 10. doi: 10.1186/s13023-025-04151-y. Online ahead of print. PMID 41366677
- [Derived] Seront E, Van Damme A, Legrand C, Bisdorff-Bresson A, Orcel P, Funck-Brentano T, Sevestre MA, Dompmartin A, Quere I, Brouillard P, Revencu N, De Bortoli M, Hammer F, Clapuyt P, Dumitriu D, Vikkula M, Boon LM. Preliminary results of the European multicentric phase III trial regarding sirolimus in slow-flow vascular malformations. JCI Insight. 2023 Nov 8;8(21):e173095. doi: 10.1172/jci.insight.173095. PMID 37937645